CLINICAL TRIAL: NCT02902406
Title: Validation of DNA Methylation Biomarkers for Oral Cancer Detection-Follow up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201601034RINB
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2016-09

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- normal oral mucosa
- oral precancerous lesion or oral cancer

SUMMARY:
This is a follow up study which aims to evaluate the correlation between several methylated genes (potential biomarkers) and oral cancers. A prospective case control trial is designed with sample size of at least 300 cases with estimated 200 subjects with precancerous lesion or oral cancer, and 100 subjects with normal oral mucosa. This study is approved by the National Taiwan University Hospital Research Ethics Committee. After signing the informed consent, all subjects will receive an intraoral examination and followed by epithelial cells collection with oral swab. The gDNA will be extracted from the oral swab collected cells and followed by bisulfite conversion procedures. Subsequently, bisulfite converted DNA will be subjected to methylated gene detection by Real-Time PCR. The methylation index (clinical sensitivity and specificity) of oral cancer related genes will be evaluated. For diagnosis confirmation, photos and biopsy specimens will be taken upon observation of abnormal lesion.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age over 20.
* Subjects with oral mucosal findings (normal, oral mucosal lichen planus, precancerous lesion, and oral cancer) or subjects who have involved in the previous study (NCT01945697).
* Subjects agrees to sign the informed consent form.

Exclusion Criteria:

* Pregnant woman.
* Subject disagrees to sign the informed consent form.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients come to the Department of Dentistry of National Taiwan University Hospital for oral health care or treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-04-18 (Actual); Primary Completion 2019-04-17 (Estimated)

PRIMARY OUTCOMES:
DNA methylation | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dentistry National Taiwan University Hospital, Taipei, Taiwan